CLINICAL TRIAL: NCT00257127
Title: Evaluation of Immunologic Memory Following Pneumococcal, Hepatitis B, and Measles Vaccination in HIV Infected Children Treated With Highly Active Antiretroviral Therapy (HAART)
Brief Title: Immune System Function Following Vaccination in HIV Infected Children Taking Anti-HIV Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1061s; 10132 (Registry Identifier: DAIDS ES Registry Number); PACTG P1061s
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccination
MeSH Terms: conditions — HIV Infections | interventions — Pneumococcal Vaccines; Hepatitis B Vaccines; Measles-Mumps-Rubella Vaccine

ARMS (2):
- 1 (Experimental): Patients will receive PCV, HBV, and MMR at study entry
  Interventions: Biological: Pneumococcal 7-valent conjugate vaccine; Biological: Hepatitis B vaccine; Biological: Measles, mumps, and rubella virus vaccine, live
- 2 (Experimental): Patients will receive PPV, HBV, and MMR at study entry
  Interventions: Biological: Pneumococcal polysaccharide vaccine; Biological: Hepatitis B vaccine; Biological: Measles, mumps, and rubella virus vaccine, live

INTERVENTIONS:
Biological: Pneumococcal 7-valent conjugate vaccine — 0.5 mL administered intramuscularly
  Other Names: PCV
  Arms: 1
Biological: Pneumococcal polysaccharide vaccine — 0.5 mL administered intramuscularly
  Other Names: PPV
  Arms: 2
Biological: Hepatitis B vaccine — 0.5 mL administered intramuscularly
  Other Names: HBV
Biological: Measles, mumps, and rubella virus vaccine, live — 0.5 mL administered subcutaneously
  Other Names: MMR

SUMMARY:
The purpose of this study is to determine immune system function following vaccination in HIV-infected children currently taking anti-HIV drugs. To test the effectiveness of prior vaccination, patients in this study will receive booster shots of one of two pneumococcal vaccines, a hepatitis B vaccine, and a measles vaccine.

DETAILED DESCRIPTION:
With their immunocompromised status, HIV-infected children are at especially high risk for opportunistic infections, including infection by Streptococcus pneumoniae, hepatitis B, and measles. In PACTG P1024, HIV-infected children taking highly active antiretroviral therapy (HAART) received 2 doses of the pneumococcal conjugate vaccine (PCV), 1 dose of the pneumococcal polysaccharide vaccine (PPV), and booster shots of the hepatitis B vaccine (HBV) and measles, mumps, and rubella vaccine (MMR). Early responses to these vaccinations were favorable, but with declining antibody responses within the 18 months after vaccination. It is unknown if additional booster vaccinations in these children will result in a protective immunologic memory upon re-exposure to these pathogens. This study will determine whether HIV-infected children on HAART have evidence of specific immunologic memory 3 to 4 years after vaccination in PACTG P1024.

Patients will be randomly assigned to receive PCV or PPV at study entry. All eligible patients will also receive HBV and MMR at study entry. Patients will be monitored in the clinic for 1 hour after vaccination for any adverse effects. Study staff will contact patients by phone around Day 3 after study entry to ask patients if they have experienced any adverse effects to the vaccinations; patients who received MMR at study entry will be contacted again around Day 21. Some patients may be asked to return to the clinic for further evaluation if they experience side effects.

There will be study visits at study entry and Days 7 and 28. Medical history, a physical exam, blood collection, and an assessment of HIV-related symptoms will occur at all visits. HAART will not be provided by this study.

ELIGIBILITY:
Inclusion Criteria:

* Completed the 96-week initial study period of PACTG P1024 and had enrolled into that study between June 1, 2001 and March 31, 2002
* Fulfilled PACTG P1024's definition of HAART (taking 3 or more antiretrovirals [ARVs] from at least 2 of the available therapeutic drug classes) during PACTG P1024's vaccination period (Weeks 0 to 24). Patients who were taking 3 nucleoside reverse transcriptase inhibitors during that period without a non-nucleoside reverse transcriptase inhibitor or a protease inhibitor (PI) are not eligible for this study. Nontherapeutic boosting doses of ritonavir used in ritonavir-boosted PI regimens are not counted as separate ARVs.
* Stable ARV regimen in the 4 weeks prior to study entry
* No changes anticipated to current ARV regimen during this study
* Willing to complete all study vaccinations and evaluations
* Willing to use acceptable forms of contraception, if applicable
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Abnormal blood or chemistry values on most recent laboratory tests. More information on this criterion can be found in the protocol.
* Received PCV, HBV, PPV, or MMR vaccines during PACTG P1024 in a sequence other than specified in PACTG P1024
* Received one or more doses of each of PCV, PPV, MMR, or HBV vaccines since the end of PACTG P1024's vaccination period
* Previous Grade 3 or higher adverse events or allergic reactions judged to be possibly or definitely related to the PCV, PPV, MMR, or HBV vaccines
* Received any killed vaccine within the 4 weeks prior to study entry
* Received any live vaccine within the 6 weeks prior to study entry
* Planning to receive any killed or live vaccine other than study vaccines between the first and third study visits
* Presence of an underlying condition that contraindicates use of any of the study vaccines. Patients who have a CD4% less than 15% will not be given the MMR vaccine, but such patients will not be excluded from this study.
* Current immunomodulatory therapy, including IL-2, any interferon product, GM-CSF, or thalidomide. Patients taking G-CSF or erythropoietin are not excluded.
* Anticipated need for immunomodulatory treatment during this study
* Any intramuscular immune globulin product within the 6 months prior to study entry
* Intravenous immune globulin within the 11 months prior to study entry
* Platelets or plasma products within the 7 months prior to study entry
* Anticipated need for immune globulin products during this study
* Current systemic immunosuppressive therapy, including the equivalent of 1 mg/kg/day or greater of prednisone in the 2 weeks prior to study entry. Patients using inhaled corticosteroids only are not excluded from this study. More information on this criterion can be found in the protocol.
* Anticipated need for systemic immunosuppressive therapy during this study
* Other known or suspected diseases of the immune system
* Cancer in the 3 months prior to study entry or treatment for cancer within the 3 months prior to study entry
* Other acute or chronic medical or surgical conditions or contraindications that, in the opinion of the investigator, may interfere with the study
* Known bleeding disorder
* Any Grade 2 or higher clinical toxicity at study screening. More information on this criterion can be found in the protocol.
* Require certain medications
* Pregnancy

Ages: 6 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2006-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Grade 3 or greater hematologic and chemistry laboratory values, signs, or symptoms not present, as specified by the protocol | At study entry

SECONDARY OUTCOMES:
Seropositivity, as determined by antibody levels | At study entry and Days 7 and 28
Immunologic memory, as determined by primary and secondary responses, antibody levels, and additional measures of immunologic memory | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Abzug, MD, Study Chair — The Children's Hospital, Denver, CO
Locations (26):
- United States (24):
  - UAB, Dept. of Ped., Div. of Infectious Diseases, Birmingham, Alabama
  - Usc La Nichd Crs, Alhambra, California
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - UCSD Mother-Child-Adolescent Program CRS, San Diego, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida College of Medicine-Dept of Peds, Div. of Immunology, Infectious Diseases & Allergy, Gainesville, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Children's Hosp., New Orleans, Louisiana
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Metropolitan Hosp. Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
- Puerto Rico (2):
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Obaro SK, Pugatch D, Luzuriaga K. Immunogenicity and efficacy of childhood vaccines in HIV-1-infected children. Lancet Infect Dis. 2004 Aug;4(8):510-8. doi: 10.1016/S1473-3099(04)01106-5. PMID 15288824
- [Derived] Abzug MJ, Song LY, Levin MJ, Nachman SA, Borkowsky W, Pelton SI; International Maternal Pediatric Adolescent AIDS Clinical Trials Group P1024 and P1061s Protocol Teams. Antibody persistence and immunologic memory after sequential pneumococcal conjugate and polysaccharide vaccination in HIV-infected children on highly active antiretroviral therapy. Vaccine. 2013 Oct 1;31(42):4782-90. doi: 10.1016/j.vaccine.2013.08.002. Epub 2013 Aug 14. PMID 23954381
- See also: Click here for more information about PACTG P1024 — http://www.clinicaltrials.gov/ct/show/NCT00013871